CLINICAL TRIAL: NCT02971488
Title: The Impact on Linkage-to-care of an Alternative Hepatitis C Screening Method in PWID
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Infanta Leonor (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Fundacion SEIMC-GESIDA (Other)
Responsible Party: Principal Investigator, Pablo Ryan, Principal Investigator, Hospital Universitario Infanta Leonor
Other Study IDs: HUIL 15/03
Record Dates: First submitted 2016-10-13; First posted 2016-11-23 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-08

CONDITIONS: Hepatitis C; Drug Users; Harm Reduction; HIV
Keywords: Hepatitis C; PWID; Linkage-to-care
MeSH Terms: conditions — Hepatitis C; Drug Misuse; Harm Reduction | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Samples were collected in DBS and sent to National Centre of Microbiology
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Persons who inject drugs (PWID): The study population comprises persons who visit the Cañada Real Galiana shantytown on the outskirts of Madrid, where 90% of illegal drugs in the region are sold and consumed.
  Interventions: Other: Screening for HCV in PWID and Linkage-To-Care

INTERVENTIONS:
Other: Screening for HCV in PWID and Linkage-To-Care — Screening, diagnosis and treatment of HCV in PWID, will be part of a harm reduction strategy.
  Treatment of HCV infected PWID will be delivered in a multidisciplinary care setting with services to reduce the risk of reinfection and for management of the common social and psychiatric comorbidities in this population.

SUMMARY:
Screening, diagnosis and treatment of HCV in PWID, should be part of a harm reduction strategy. Treatment of HCV infected PWID should be delivered in a multidisciplinary care setting with services to reduce the risk of reinfection and for management of the common social and psychiatric comorbidities in this population. More frequent diagnosis, new methods that prevent loss of tracking, and access to antiviral treatment are all strategies that must be implemented jointly if the prevalence of HCV infection in our setting is to be reduced.

ELIGIBILITY:
Inclusion Criteria:

* PWID
* >18 years of age
* Signed consent form

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population comprises persons who visit the Cañada Real Galiana shantytown on the outskirts of Madrid, where 90% of illegal drugs in the region are sold and consumed. It is estimated that between 4000 and 6000 people per day visit the shantytown for their dose. The regional government's Anti-Drug Agency has a mobile HRU operating daily in the area. The unit provides screening tests to anyone who is willing to take them, regardless of whether they are already aware of their serological status or not. Screening includes education on prevention of HCV infection and other transmissible diseases.
Sampling Method: Non-Probability Sample
Enrollment: 529 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-05-10 (Actual)

IPD SHARING:
Plan to Share IPD: No
not shared in public

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Patients: All the patients in the study
Period: Overall Study
Arm/Group | Total Patients
Started | 529
Completed | 529
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Persons Who Inject Drugs (PWID): The study population comprises persons who visit the Cañada Real Galiana shantytown on the outskirts of Madrid, where 90% of illegal drugs in the region are sold and consumed.
  Screening for hepatitis C virus (HCV) in PWID and Linkage-To-Care: Screening, diagnosis and treatment of HCV in PWID, will be part of a harm reduction strategy.
  Treatment of HCV infected PWID will be delivered in a multidisciplinary care setting with services to reduce the risk of reinfection and for management of the common social and psychiatric comorbidities in this population.
Arm/Group | Persons Who Inject Drugs (PWID)
Number analyzed (Participants) | 529
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 42 [35 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109
  Male | 420
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Spain | 529
Homelessness [Count of Participants; unit: Participants] — Participants who were homeless
  Participants | 105
Spanish born [Count of Participants; unit: Participants] — Participants who were born in Spain
  Participants | 419
Type of drug used [Count of Participants; unit: Participants]
  Heroine | 412
  Cocaine | 476
  Alcohol | 50
Current way of administration of drug [Count of Participants; unit: Participants]
  Injected | 177
  Smoked | 432
  Snorted | 135
Retained in care [Count of Participants; unit: Participants] — Participants who have access or are followed up in a healthcare center (addiction center, harm reduction unit, mental health center...)
  Participants | 449
Never tested [Count of Participants; unit: Participants] — Participants who had never been tested for HIV or HCV before study inclusion
  Participants
    Never tested for HIV | 57
    Never tested for HCV | 55
Participants with Opioid Substitute Treatment (OST) [Count of Participants; unit: Participants] | 142
Stable partner [Count of Participants; unit: Participants] — Participants who currently have a stable partner
  Participants | 204

OUTCOME MEASURES:

1. Primary Outcome: Percentage of HCV Infected Paticipants Whom Result of the Test Was Delivered to
Description: Percentage of participants who had a positive HCV test and results of the test was delivered to them.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Participatnts With an Active HCV Infection: Participants who had tested positive for hepatitis C (Positive PCR).
Arm/Group | Participatnts With an Active HCV Infection
Number analyzed (Participants) | 122
Participants | 101

2. Primary Outcome: Percentage of Participants Who Were Evaluated at a HCV Clinic.
Description: Evaluation of the effectiveness of the intervention. Subjects who had a positive result in the screening performed in Cañada Real Galiana will be contacted and offered the possibility of referral to HUIL, where they will have access to standard confirmation tests. Here, test accuracy will be evaluated at population level. Patients will have access to HCV treatment and will be followed for assessment of the impact of the program on patients' health (appointment in health centers, percentage of treated patients, and the percentage of virological response).
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- HCV Infected Patients: Those with an active HCV infection
Arm/Group | HCV Infected Patients
Number analyzed (Participants) | 122
Participants | 63

3. Primary Outcome: Percentage of Participants Who Started HCV Antiviral Therapy.
Description: as for outcome 2
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | HCV Infected Patients
Number analyzed (Participants) | 122
Participants | 52

4. Primary Outcome: Percentage of Participants Who Achieved a Sustained Virological Response (SVR)
Description: as for outcome 2
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Patients Who Started HCV Therapy: HCV infected Patients who started treatment with antivirals
Arm/Group | HCV Infected Patients | Patients Who Started HCV Therapy
Number analyzed (Participants) | 122 | 52
Participants | 38 | 38

5. Secondary Outcome: Percentage of Participants With Active HCV in Screened Population
Description: Screening for HCV using dried blood samples on WhatmanTM cards in subjects from Cañada Real based on the results of the laboratory tests performed in phase I. The percentage of active HCV infections will be calculated from the total population of active drug addicts screened.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Total Patients
Number analyzed (Participants) | 529
Participants | 122

6. Secondary Outcome: Prevalence of Other Chronic Viral Infections in the Population Screened
Description: Other viruses (HIV, HBV, HDV) using dried blood samples on WhatmanTM cards in subjects from Cañada Real based will be analysed. The prevalence of these infections will be calculated base on the total screened population.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Total Patients
Number analyzed (Participants) | 529
Participants
  HIV infection | 35
  Hepatitis B Antigen | 23
  Hepatitis D | 2

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Total Patients
All-Cause Mortality (participants affected / at risk) | 0/529
Serious Adverse Events (participants affected / at risk) | 0/529
Other Adverse Events (participants affected / at risk) | 0/529

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-20): https://cdn.clinicaltrials.gov/large-docs/88/NCT02971488/Prot_SAP_000.pdf